CLINICAL TRIAL: NCT05850611
Title: The Effect of Combination Therapy of Oral Methylene Blue and Platelet-rich Plasma-fibrin Glue in Patients With Non-healing Diabetic Foot Ulcer: a Pilot Study
Brief Title: The Effect of Combination Therapy of Oral MB and PRP-FG in Patients With Non-healing Diabetic Foot Ulcer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Daryoush Hamidi Alamdari, PhD, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRCT20191228045924N3
Record Dates: First submitted 2023-03-06; First posted 2023-05-09 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Foot Ulcers; Diabetic Wound
Keywords: Platelet-Rich Plasma-Fibrin Glue; DFU; Methylene blue; Non-healing Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Methylene Blue; Milk

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methylene Blue (Experimental): The first intervention group (group A) includes diabetic patients with chronic foot ulcers who, despite common treatments, will be undergone oral methylene blue intervention (70 mg in 200 ml of milk) for 4 weeks.
  Interventions: Drug: Methylene Blue
- Milk (control) (Experimental): Patients with non-healing Diabetic Foot Ulcers only will receive 200 ml of milk for 4 weeks.
  Interventions: Other: Milk (control)
- Methylene Blue and Platelet-Rich Plasma-Fibrin Glue (Experimental): Patients with non-healing Diabetic Foot Ulcers will treat with PRP-Fibrin-Glue plus oral methylene blue (70 mg in 200 ml of milk) for 4 weeks.
  Interventions: Drug: Methylene Blue and Platelet-Rich Plasma-Fibrin Glue
- Milk and Platelet-Rich Plasma-Fibrin Glue (control) (Experimental): Patients with non-healing Diabetic Foot Ulcers will be treated with PRP-Fibrin-Glue and 200 ml of milk for 4 weeks.
  Interventions: Other: Milk and Platelet-Rich Plasma-Fibrin Glue (control)

INTERVENTIONS:
Drug: Methylene Blue — The first intervention group includes diabetic patients with chronic foot ulcers who, despite common treatments, will be undergone oral methylene blue intervention for 4 weeks.
  Other Names: Methylthioninium chloride
  Arms: Methylene Blue
Other: Milk (control) — Group B will receive 200 ml of milk for 4 weeks.
  Other Names: Placebo
  Arms: Milk (control)
Drug: Methylene Blue and Platelet-Rich Plasma-Fibrin Glue — Group C will be undergone synergistic 4-week treatment with oral methylene blue and fibrin glue.
  Other Names: Methylthioninium chloride and PRP-Fibrin Glue
  Arms: Methylene Blue and Platelet-Rich Plasma-Fibrin Glue
Other: Milk and Platelet-Rich Plasma-Fibrin Glue (control) — Group D will be treated only with fibrin glue and 200 ml of milk for 4 weeks.
  Other Names: Placebo
  Arms: Milk and Platelet-Rich Plasma-Fibrin Glue (control)

SUMMARY:
The aim of this study is to evaluate the chance of non-healing diabetic foot ulcers repair by improving the condition of lack of oxygen or hypoxia in the wound area caused by diabetes using methylene blue along with the use of platelet-rich plasma-fibrin glue as an effective treatment for wound healing.

DETAILED DESCRIPTION:
The current study assesses the effects of methylene blue along with the use of platelet-rich plasma-fibrin glue on wound healing in patients with nonhealing diabetic foot ulcers (non-healing DFU). This randomized controlled trial is performed on 20 patients with non-healing DFU. Patients were treated with PRP-FG dressing plus 200 ml of oral methylene blue dissolved in milk(intervention group) or PRP-FG dressing plus placebo (200 ml of milk) (control group) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a Diabetic ulcer grade II and IV based on Wagner's classification on the sole, medial, or lateral part of the foot (including all surfaces of the toes)
* Having a single ulcer on the feet and extremities (toes, soles, heels) with no significant reduction in ulcer size (<20%) despite the use of best treatment methods for at least four weeks
* If there is more than one non-healing wound, choose the largest wound
* The size of the wound surface (length × width) between 2 cm2 and 20 cm2
* No smoking, alcohol, and drug addiction based on the patient's self-report
* Not taking drugs that may interfere with wound healing, such as Corticosteroids, immunosuppressants, and cytotoxic agents
* Not having a concurrent chronic disease that may cause problems in wound healing, such as cancers, vasculitis, no history of known severe kidney, liver, and heart disease, such as liver cirrhosis, active hepatitis, dialysis, etc.
* Not taking antidepressants
* Insensitivity to milk lactose
* Not having Glucose 6-phosphate dehydrogenase (G6PD) deficiency
* Confirmed, informed, signed consent form
* Ankle Brachial Index (ABI) higher than or equal to 0.7

Exclusion Criteria:

* Do not be treated with methylene blue
* The confirmed presence of osteomyelitis, or if there is suspicion of osteomyelitis
* The subject is pregnant or intends to become pregnant during the test period
* The patient is known to have mental, developmental, physical, and emotional disorders
* The occurrence of certain medical conditions
* The presence of a wound with a clear and severe infection, which is characterized by significant purulent secretions or extensive cellulitis, or gangrene requiring amputation
* Evidence of venous, ischemic, neurotrophic ulcers (numbness, tingling, lack of Achilles tendon reflex) and traumatic wounds in the patient
* Failure to refer the patient more than two times to the mentioned center for follow-up and dressing change
* Hypersensitivity reaction to methylene blue
* Platelet count less than 100,000
* The patient's lack of consent to continue cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-09-21 (Estimated)

PRIMARY OUTCOMES:
The healing rate of the ulcer | 4 weeks
  Measurement of wound area with a ruler
Wound Size | 4 weeks
  Wound size will be measured with a ruler for length, and width as well as with digital imaging. Wound size will be assessed in digital images taken of the wound.

SECONDARY OUTCOMES:
TcPO2 at baseline and after the intervention | 4 weeks
  Transcutaneous oxygen tension (TcpO2) provides information about blood perfusion in the tissue immediately below the skin. (blood pressure, measured in millimeters of mercury (mmHg))
Oxygen saturation at baseline and after the intervention | 4 weeks
  Blood must contain a normal concentration of hemoglobin. that hemoglobin must be >95 % saturated with oxygen in arterial blood (sO2(a) >95 %)
Blood pressure (systolic and diastolic) | 4 weeks
  The pressure of the blood in the circulatory system
The resting systolic toe pressure (TP) at baseline and after the intervention | 4 weeks
  The toe cuff with the sphygmomanometer is slowly inflated until the waveform flattens (generally between 150-200 mmHg), then is inflated a further 20 mmHg. The cuff is slowly released at a rate of 2-5mmHg per second. The first regular cyclical waveform is considered the toe systolic pressure.
Serum IL-1β levels at baseline and after the intervention | 4 weeks
  Analysis of serum interleukin-1β levels
Serum MCP-1 levels at baseline and after the intervention | 4 weeks
  Analysis of serum monocyte chemoattractant protein-1 (MCP-1) levels
Serum TNF-α levels at baseline and after the intervention | 4 weeks
  Analysis of serum tumor necrosis factor α (TNFα) levels
Serum IL-6 levels at baseline and after the intervention | 4 weeks
  Analysis of serum interleukin-6 (IL-6) levels
Serum HIF-1α levels at baseline and after the intervention | 4 weeks
  Analysis of serum hypoxia-inducible factor 1-alpha (HIF-1α) levels
Serum FBS levels at baseline and after the intervention | 4 weeks
  Analysis of serum fasting blood sugar (FBS ) levels
Serum Insulin levels at baseline and after the intervention | 4 weeks
  Analysis of Insulin levels
Lipid Profile at baseline and after the intervention | 4 weeks
  Serum Triglyceride, Cholesterol, HDL, LDL, VLDL
Serum Urea at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Creatinine at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum total bilirubin at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Vitamin D levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
HbA1c at baseline and after the intervention | 4 weeks
  Glycated hemoglobin
Serum Albumin (Alb) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Uric Acid levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Homocysteine levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum ALT (alanine transaminase) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum AST (Aspartate Transferase) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum ALP (alkaline phosphatase) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Met Hemoglobin levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Hemoglobin (Hgb, Hb) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum white blood cells (WBCs) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum total Lymphocyte levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Platelet count at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Nitric oxide blood at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum lactate dehydrogenase (LDH) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum Erythrocyte Sedimentation Rate (ESR) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Serum C-Reactive Protein (CRP) levels at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method
Neutrophils count at baseline and after the intervention | 4 weeks
  In a quantitative laboratory method

CONTACTS AND LOCATIONS:
Overall Officials: Daryoush Hamidi Alamdari, Ph.D, Principal Investigator — Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
All data related to the project after the unidentifiable people will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Access to data is allowed 6 months after the publication of results.
Access Criteria: The investigator's data will be available to university staff and academic institutions.